CLINICAL TRIAL: NCT05302609
Title: Phase II Study: Evaluation of SclerFIX Graft in Scleral Thinning After Exeresis of Tumors of the Ocular Surface
Brief Title: Evaluation of SclerFIX Graft in Scleral Thinning After Exeresis of Tumors of the Ocular Surface
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SclerFIX-TBF3; 2021-A02109-32 (Other: IDRCB)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Scleral Thinning
Keywords: Ocular Oncology; Tumor Exeresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SclerFIX (Experimental): Patch of umbilical cord lining membrane sutured on top of the scleral defect.
  Interventions: Biological: SclerFIX

INTERVENTIONS:
Biological: SclerFIX — Chemically-treated, viro-inactivated, freeze-dried and irradiated umbilical cord lining membrane allograft used as substitute for scleral graft in reinforcement of scleral thinning.

SUMMARY:
The purpose of this open, multicenter phase II trial is to confirm the tolerance and evaluate the efficacy of the SclerFIX product, an allograft of umbilical cord lining membrane, in reinforcement of scleral thinning in patients who underwent eye tumor exeresis.

DETAILED DESCRIPTION:
As scleral graft is forbidden in France, it cannot be used to reinforce the sclera. This study investigational product, SclerFIX, was developed to substitute scleral grafts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80 years.
* Patients with risk of perforation or deep loss of substance during surgical removal of a tumor of the ocular surface.
* Patient with loss of substance < 3cm2.
* Patient able to understand, sign and date the informed consent form.
* Patient who is a member or a beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman or woman of childbearing age without effective contraception.
* Patients with uncontrolled infectious risk.
* Patient with an autoimmune disease.
* Person deprived of liberty by a judicial or administrative decision.
* Person under forced psychiatric care.
* Person admitted to a health or social institution for purposes other than the research.
* Adult subjected to a legal protection measure or unable to express his / her consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Rate of tectonic success of the graft at 3 months | 3 months
  The graft will be considered successful at 3 months if the curvature of the eye is respected without thinning, i.e., in the absence of edema, ulceration and loss of substance (thickness of the grafted area/thickness of the adjacent surface > 80%). The scleral thickness will be determined from images obtained by optical coherence tomography (OCT).

SECONDARY OUTCOMES:
Absence of inflammatory reactions and good local tolerance of the implant | 15 days, 1 month, 3 months
  Composite score evaluating the presence of local reactions (edema, redness, vascularization, discharge) and of ulceration, pain and foreign body sensation (0: excellent local tolerance, 46: worst possible local tolerance)
Evaluation of the visual acuity | 15 days, 1 month, 3 months
  Scoring of blurred and poor vision (0: never, 4: all the time)
Evaluation of the eye pressure | 15 days, 1 month, 3 months
  Measure of eye pressure using a tonometer

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Hôpital Pasteur 2 - CHU de NICE, Nice

IPD SHARING:
Plan to Share IPD: No